CLINICAL TRIAL: NCT04792346
Title: a Feasibility Study of Accelerated Hypofractionated Radiotherapy in Node Positive Breast Cancer Patients Treated With Surgery
Brief Title: Ten Fraction Adjuvant Hypofractionated Radiotherapy in Node Positive Breast Cancer
Acronym: HIPOMAMMLINF
Status: Completed | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Giuseppe Sanguineti (Unknown); Silvia Takanen (Unknown); Serena Nucciarelli (Unknown); Francesco Rulli (Unknown); Maria Papale (Unknown); Valeria Landoni (Unknown); Mauro Caterino (Unknown); Diana Giannarelli (Unknown); Ilaria Farina (Unknown); Paola Franzoso (Unknown)
Responsible Party: Principal Investigator, Paola Pinnaro, Doctor, Regina Elena Cancer Institute
Other Study IDs: RS618/14(1611)
Record Dates: First submitted 2021-03-02; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer
Keywords: hypofractionated RT; cosmetic outcome; locoregional treatment
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: breast/chest wall radiotherapy — 34 Gy/10 fxs/2 wks to the whole breast/chest wall and locoregional lymph nodes; an optional single fraction 8 Gy boost was administered with electrons to the tumor bed in patients undergoing conservative surgery

SUMMARY:
Post-operative loco-regional (LR) hypofractionated radiotherapy (Hypo-RT) is an attractive approach in locally advanced breast cancer (LABC).

DETAILED DESCRIPTION:
The present is a single arm phase II study assessing toxicity levels after 34 Gy/10 fxs/2 wks to the whole breast/chest wall and to the draining lymph nodes; an optional single fraction 8 Gy boost was administered with electrons to the tumor bed in patients who had undergone conservative surgery. Both acute (CTCAE v4.0) and late (LENT/SOMA) toxicity were collected. All pts but those who underwent mastectomy without reconstruction or with temporary expander were also asked to rate their cosmetic outcome according to the Harvard. Toxicity was assessed weekly during RT and then at each follow-up examination (1, 3, 6 months and then yearly).

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by invasive breast cancer who underwent conservative breast surgery or mastectomy and axillary dissection, followed by post operative radiotherapy at the level of the breast/chest wall, and of the supraclavicular, third axillary level +/- internal mammary chain nodes.
* pT1-3 disease pN1-2, cT1-3 disease if neoadjuvant chemotherapy , cN + cytologically and/or histologically assessed;
* ECOG Performance status ≤2;
* histologically negative surgical margins
* no distant metastases
* no prior chest radiotherapy
* life expectancy ≥ 5 years
* no prior cancer

Exclusion Criteria:

* Non-epithelial breast cancer (sarcoma, lymphoma etc.)
* Metastases at the level of the internal chain mammary and / or supra-clavicular lymph nodes histologically assessed
* pT4 neoplasms or inflammatory breast carcinoma
* Distant metastasis
* Concomitant chemotherapy
* history of prior controlateral breast tumor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population included breast cancer patients with nodal involvement who underwent conservative surgery or mastectomy, followed by post operative locoregional radiotherapy after conservative surgery or mastectomy.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
acute toxicity assessment | 60 months
  rate of acute toxicity according to CTCAE v4.0 scale

SECONDARY OUTCOMES:
to evaluate late toxicity | 60 months
  rate of late to according to soma lent scale

CONTACTS AND LOCATIONS:
Overall Officials: Paola Pinnaro, Principal Investigator — IFO
Locations (1):
- Regina Elena National Cancer Institute, Rome, Italy

IPD SHARING:
Plan to Share IPD: No